CLINICAL TRIAL: NCT03741556
Title: Recovery Following Ankle Fracture Reported by Patient Report Outcome
Brief Title: Prognostic Factors Following Ankle Fractures
Status: Completed | Type: Observational
Sponsor: Sygehus Lillebaelt (Other)
Collaborators: Kolding Sygehus (Other)
Responsible Party: Principal Investigator, per hviid gundtoft, Principal Investigator, Senior House Officer, PhD, Sygehus Lillebaelt
Other Study IDs: Ver2
Record Dates: First submitted 2018-11-06; First posted 2018-11-15 (Actual); Last update posted 2023-08-07 (Actual); Status verified 2023-08

CONDITIONS: Ankle Fractures
MeSH Terms: conditions — Ankle Fractures

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: questionaire — a questionaire is sent to each participans

SUMMARY:
Ankel fractures is a common fracture. Most patients experience that the regain normal range of motions and limited pain within the first 6 months following ankel fracture, but not all. The aim of the study is to determine if any prognostic factors is associated with a worse outcome.

DETAILED DESCRIPTION:
Aim of study:

To identify prognostic factors associated with a worse outcome following ankle fractures.

Method:

All operated or non-operated ankle fractures in a period of one year from three different hospitals will be included. The following data will be recorded:

Civil registration number, age, rupture of the syndesmosis, use of alcohol, smoking, diabetes, characteristics of the ankle fracture (AO classification), type of treatment and complications.

Study participants will at time of diagnosis and 6, 12, 52 and 104 weeks following the injury received a questionaire with Manchester foot and ankle questionnaire (MOXFQ), Self-reported foot and ankle questionnaire (SEFAS), Olerud Molander Ankle Score (OMAS) and Forgotten Joint Score (FJS).

Which of the questionaire that should be used in the study will be determined when the questionaires have been compared in a different study.

ELIGIBILITY:
Inclusion Criteria:

* All patients with ankle fracture.

Exclusion Criteria:

* age below 18 years
* patients who do not speak or understand danish
* mental disable patients

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All patients with an ankle fracture, treated either with an operation or non-operative in one of three hospitals
Sampling Method: Non-Probability Sample
Enrollment: 160 (Actual)
Dates: Start 2018-11-07 (Actual); Primary Completion 2020-07-01 (Actual); Study Completion 2022-10-01 (Actual)

PRIMARY OUTCOMES:
Manchester foot and ankle questionnaire (MOXFQ) | 2 years
  Manchester foot and ankle questionnaire (MOXFQ) a Patient reported outcome measure. The MOXFQ contains 16 items, each with five response options, comprising three dimensions: walking/standing problems (seven items), foot pain (five items), and issues related to social interaction (four items), including feelings of self consciousness about foot/footwear appearance. Responses are each scored from 0 to 4, with 4 representing the most severe response. Item responses are summed to give a score from 0-100, with higher score representing the worse possible
Self-reported foot and ankle questionnaire (SEFAS) | 2 years
  The Self-reported foot and ankle questionnaire (SEFAS) comprises twelve items relating to pain, limping, swelling, use of orthotics and walking. Response scales vary from 1 to 5, 1 being the most severe response. Item responses are summed to give a score from 12-60, with higher scores representing the best possible.
Olerud Molander Ankle Score (OMAS) | 2 years
  The Olerud Molander Ankle Score (OMAS) comprises nine items relating to symptoms, physical function and daily activities. The response scales vary from binary to five-points with clinical scoring that reflects the level of disability for individual items. Item responses are summed to give a score from 0 to 100 with higher scores representing the best possible
Forgotten Joint Score (FJS) | 2 years
  The forgotten Joint Score (FJS) is a 12-item questionnaire concerning the participiants awareness of their artificial joint during ADL. For each question, the participant can choose between 6 response options: never, almost never, seldom, sometimes, mostly, or not relevant for me. All responses are summed from 0-4 with a total score from 0-100 with higher scores representing the worse possible

SECONDARY OUTCOMES:
EQ5D-3L | 2 years
  The EQ5D-3L is a generic PROM and does not specifically address foot and ankle disability. The EQ-5D-3L includes five items with a three-point response scale which are scored to give a single index, with 0 representing the worse possible disability. It also includes a visual analoug scale (VAS) to assess general health, ranging from 0-100, with 0 representing the worse possible health state

CONTACTS AND LOCATIONS:
Locations (3):
- Denmark (3):
  - Amager Hvidovre Hospital, Copenhagen
  - Sygehus Lillebaelt, Kolding
  - Odense University Hospital, Odense

IPD SHARING:
Plan to Share IPD: No
We do not plan to share the data.